CLINICAL TRIAL: NCT06162221
Title: A Platform Study of RAS(ON) Inhibitors in Patients With RAS-Mutated Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study of RAS(ON) Inhibitors in Patients With Advanced RAS-mutated NSCLC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Revolution Medicines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC-LUNG-101
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-06

CONDITIONS: Non-Small Cell Lung Cancer, NSCLC; KRAS, NRAS, HRAS-mutated NSCLC; KRAS G12C-mutated Solid Tumors, Lung Cancer; Lung Cancer Stage IV, Advanced Solid Tumor, Cancer; RAS G12D-mutated NSCLC
Keywords: NSCLC; KRAS G12C; RAS Mutation; KRAS G12X; Non-Small Cell Lung Cancer; Lung Cancer; Lung Cancer Stage IV; Advanced Solid Tumor; Cancer; RAS G12D
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasms | interventions — pembrolizumab; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Subprotocol A: KRAS G12C-Mutated Solid Tumors (Experimental): RMC-6291 (BID), RMC-6236 (QD), and Pembrolizumab (Q3W) with or without Chemotherapy (Q3W)
  Interventions: Drug: RMC-6291; Drug: RMC-6236; Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed
- Subprotocol B: RAS-mutated NSCLC (Experimental): RMC-6236 (QD) and Pembrolizumab (Q3W) with or without Chemotherapy (Q3W)
  Interventions: Drug: RMC-6236; Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed
- Subprotocol C: RAS G12D-mutated NSCLC (Experimental): RMC-9805 (QD or BID), RMC-6236 (QD), and Pembrolizumab (Q3W) with or without Chemotherapy (Q3W).
  Interventions: Drug: RMC-6236; Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: RMC-9805
- Subprotocol D: RAS G12D-mutated NSCLC (Experimental): RMC-9805 (QD)
  Interventions: Drug: RMC-9805

INTERVENTIONS:
Drug: RMC-6291 — Oral tablet
  Arms: Subprotocol A: KRAS G12C-Mutated Solid Tumors
Drug: RMC-6236 — Oral tablet
  Arms: Subprotocol A: KRAS G12C-Mutated Solid Tumors; Subprotocol B: RAS-mutated NSCLC; Subprotocol C: RAS G12D-mutated NSCLC
Drug: Pembrolizumab — IV Infusion
  Arms: Subprotocol A: KRAS G12C-Mutated Solid Tumors; Subprotocol B: RAS-mutated NSCLC; Subprotocol C: RAS G12D-mutated NSCLC
Drug: Cisplatin — IV Infusion
  Arms: Subprotocol A: KRAS G12C-Mutated Solid Tumors; Subprotocol B: RAS-mutated NSCLC; Subprotocol C: RAS G12D-mutated NSCLC
Drug: Carboplatin — IV Infusion
  Arms: Subprotocol A: KRAS G12C-Mutated Solid Tumors; Subprotocol B: RAS-mutated NSCLC; Subprotocol C: RAS G12D-mutated NSCLC
Drug: Pemetrexed — IV infusion
  Arms: Subprotocol A: KRAS G12C-Mutated Solid Tumors; Subprotocol B: RAS-mutated NSCLC; Subprotocol C: RAS G12D-mutated NSCLC
Drug: RMC-9805 — Oral Tablet
  Arms: Subprotocol C: RAS G12D-mutated NSCLC; Subprotocol D: RAS G12D-mutated NSCLC

SUMMARY:
The purpose of this platform study is to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary antitumor activity of novel RAS(ON) inhibitors as a monotherapy or combined with Standard(s) of Care (SOC) or with each other.

The first four subprotocols include the following:

Subprotocol A: RMC-6291 +/- RMC-6236 + SOC Subprotocol B: RMC-6236 + SOC Subprotocol C: RMC-9805 +/- RMC-6236 + SOC Subprotocol D: RMC-9805

DETAILED DESCRIPTION:
The platform study design allows combinations of RAS(ON) inhibitors with other anticancer agents or as a monotherapy to be evaluated in patients with RAS-mutated solid tumors with a focus on NSCLC.

This is an open-label platform Phase 1b/2 study to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary antitumor activity of novel RAS(ON) inhibitors combined with Standard of Care (SOC), or as a monotherapy and to define the Recommended Phase 2 Dose and Schedule (RP2DS). Enrollment of patients with KRAS or RAS mutations will be specified in each subprotocol.

Subprotocol A is an open-label, multicenter, Phase 1b/2 study of RMC-6291, with or without RMC-6236, in combination with pembrolizumab, with or without chemotherapy, in patients with KRAS G12C-mutated advanced solid tumors.

Subprotocol B is an open-label, multicenter, Phase1b/2 study of RMC-6236 in combination with pembrolizumab, with or without chemotherapy, in patients with RAS-mutated non-small cell lung cancer (NSCLC)

Subprotocol C is an open-label, multicenter, Phase1b/2 study of RMC-9805 with or without RMC-6236, in combination with other anticancer agents, in patients with RAS G12D-mutated non-small cell lung cancer (NSCLC)

Subprotocol D is a Phase 2, Open-label, Multicenter Study of Zoldonrasib (RMC-9805) in Previously Treated Patients with RAS G12D-Mutant Non-Small Cell Lung Cancer (NSCLC)

Subprotocols A, B, and C consist of two parts: Part 1 - Dose Exploration and Part 2 - Dose Expansion. Subprotocol D consists of only one part.

ELIGIBILITY:
Inclusion criteria:

All Patients (unless otherwise noted):

* ≥ 18 years of age
* ECOG PS is 0 to 1
* Adequate organ function as outlined by the study
* Received prior standard therapy appropriate for tumor type and stage
* Must have pathologically documented, locally advanced or metastatic KRAS G12C-mutated solid tumor malignancy (not amenable to curative surgery) (Subprotocol A)
* Must have pathologically documented, locally advanced or metastatic RAS-mutated NSCLC (Subprotocol B)
* Must have pathologically documented, locally advanced or metastatic RAS G12D-mutated NSCLC (Subprotocol C and Subprotocol D)

Exclusion criteria:

All Patients:

* Primary central nervous system (CNS) tumors
* Impaired gastrointestinal (GI) function that may significantly alter the absorption of RMC drugs
* Major surgery < 28 days of first dose
* Active or history of interstitial lung disease (ILD) or pneumonitis requiring steroids

Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Up to 5 years
  Incidence and severity of treatment-emergent Adverse Events (AEs) and serious AEs and clinically significant changes in laboratory values, ECGs and vital signs
Dose limiting toxicities | 21 days
  Number of participants with dose limiting toxicities

SECONDARY OUTCOMES:
Drug concentrations over time | Up to 21 weeks
  Observed blood concentration of each drug as applicable per subprotocol
Cmax | Up to 21 weeks
  Maximum observed blood concentration of each drug as applicable per subprotocol
Tmax | Up to 21 weeks
  Time to reach maximum blood concentration of each drug as applicable per subprotocol
AUC | Up to 21 weeks
  Area under the concentration-time curve of each drug as applicable per subprotocol
ORR | Up to 5 years
  Objective Response Rate per RECIST v1.1
DOR | Up to 5 years
  Duration of Response per RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Revolution Medicines, Study Director — Revolution Medicines
Locations (88):
- United States (26):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope - Duarte, Duarte, California
  - City of Hope - Lennar, Irvine, California
  - UC Davis, Davis Comprehensive Cancer Center, Sacramento, California
  - University of California, San Diego Moores Cancer Center, San Diego, California
  - UCSF Medical Center - Mission Bay, San Francisco, California
  - Stanford University - Stanford Cancer Institute, Stanford, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Boca Raton Clinical Research Associates, Plantation, Florida
  - Cancer Specialists of North Florida, Saint Augustine, Florida
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Cancer - Detroit (Brigitte Harris Cancer Pavilion), Detroit, Michigan
  - Intermountain Health - St. Vincent Frontier Cancer Center, Billings, Montana
  - Nebraska Cancer Specialist, Grand Island, Nebraska
  - New York University Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Clinical Research Alliance, Westbury, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Baptist Medical Center, Memphis, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology Dallas, Irving, Texas
  - NEXT Oncology Virginia, Fairfax, Virginia
- Australia (4):
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Monash Health, Clayton, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Department of Oncology, Odense
- France (14):
  - Hospices Civils de Lyon - Hôpital Louis Pradel, Bron, Auvergne-Rhône-Alpes
  - Centre Georges François Leclerc, Dijon, Bourgogne-Franche-Comté
  - CHU de Lille Institut Cœur Poumon, Lille, Hauts-de-France
  - CHU de Nantes, Nantes, Hauts-de-France
  - EDOG - Institut Bergonié, Bordeaux, Nouvelle-Aquitaine
  - Institut de Cancerologie de Ouest (ICO) - Angers, Angers
  - Ambroise-Paré Hospital, Boulogne
  - Centre François Baclesse, Caen
  - Hôpital Cochin, Paris
  - Hopital Tenon - AP-HP, Paris
  - Hopital Foch, Suresnes
  - Oncopole Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
  - Institut Curie, Paris, Île-de-France Region
- Germany (7):
  - Charite-Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
  - Uniklinik Köln, Cologne
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Thoraxklinik Heidelberg gGmbH - Universitätsklinikum Heidelberg, Heidelberg
  - Lungenfachklinik Immenhausen, Immenhausen
  - Krankenhaus Bethanien Moers, Moers
- Greece (2):
  - Henry Dunant Hospital Center, Athens
  - Thoracic General Hospital of Athens "I SOTIRIA", Athens
- Italy (7):
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST S.r.l, Meldola, Emilia-Romagna
  - Fondazione IRCCS Istituto Nazionale dei tumori, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - A.O.U. San Luigi Gonzaga-Orbassano - SCDU Oncologia Medica, Orbassano
  - Ospedale Santa Maria Delle Croci, Ravenna
  - IRCCS Instituto Nazionale tumori Ragina Elena, Rome
  - Fondazione Policlinico Universitario A Gemelli-Rome, Rome
- Netherlands (4):
  - The Netherlands Cancer Institute (NKI), Amsterdam
  - University Medical Centre Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - University Medical Center Utrecht, Utrecht
- South Korea (5):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul, Seocho-gu
  - Severance Hospital, Seoul, Seodaemun-Gu
- Spain (12):
  - Hospital Clinico San Carlos, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia, Valencia
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitari Vall D' Hebron, Barcelona
  - ICO Badalona - H.U. Germans Trias i Pujol, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Regional Universitario de Malaga - Hospital Civil, Málaga
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Fundacion Instituto Valenciano de Oncologia, Valencia
- Taiwan (5):
  - Taipei Municipal Wanfang Hospital, Taipei, Wenshan Dist
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Hospital, Liouying, Tainan
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Derived] Cregg J, Edwards AV, Chang S, Lee BJ, Knox JE, Tomlinson ACA, Marquez A, Liu Y, Freilich R, Aay N, Wang Y, Jiang L, Jiang J, Wang Z, Flagella M, Wildes D, Smith JAM, Singh M, Wang Z, Gill AL, Koltun ES. Discovery of Daraxonrasib (RMC-6236), a Potent and Orally Bioavailable RAS(ON) Multi-selective, Noncovalent Tri-complex Inhibitor for the Treatment of Patients with Multiple RAS-Addicted Cancers. J Med Chem. 2025 Mar 27;68(6):6064-6083. doi: 10.1021/acs.jmedchem.4c02314. Epub 2025 Mar 8. PMID 40056080